CLINICAL TRIAL: NCT05315141
Title: Multicenter Cohort Study of ANCA-associated Small Vasculitis in Hunan Province of China
Brief Title: Multicenter Cohort Study of AAV in Hunan of China
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Hunan Provincial People's Hospital (Other); Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Xiangcheng Xiao, Professor, Xiangya Hospital of Central South University
Other Study IDs: 202108374
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: ANCA Associated Vasculitis
Keywords: ANCA Associated Vasculitis; ESRD; Outcome
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Xiangya Hospital
  Interventions: Other: No Intervention
- The Second Xiangya Hospital
  Interventions: Other: No Intervention
- The Third Xiangya Hospital
  Interventions: Other: No Intervention
- Hunan Provincial People's Hospital
  Interventions: Other: No Intervention
- Xiangtan Central Hospital
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This study aimed to explore the incidence of Anti-neutrophil cytoplasmic antibody (ANCA）-associated vasculitis (AAV) progression and its association with adverse consequences. It will enroll approximately 500 AAV patients in Hunan province of China and follow-up for at least 5 years. Demographic characteristics, clinical and laboratory data will be collected at baseline and every follow-up. The principal clinical outcomes of the study consist of end stage renal disease (ESRD) and death.

DETAILED DESCRIPTION:
The study is a multicenter prospective cohort study, aimed to explore the incidence of AAV and its progression and association with adverse consequences. The study will establish a baseline cohort of 500 AAV patients in Hunan province of China. The follow-up will be conducted for at least 5 years until death or starting renal replacement therapy or dropout. Their demographic characteristics, clinical data, laboratory and imaging examinations will be collected at baseline and every follow-up.

The baseline visit includes the following items: detailed demographics, medical and family history, medication history, health behaviors, physical activity, and anthropometric measures. The laboratory parameters of chemistry test. After the baseline visit, participants will return annually for follow-up visits and evaluation. The evaluating items of follow-up visits are similar to the baseline visit, and sample collection.

The principal clinical outcomes of the study can be broadly categorized as end stage renal disease and death. Death is further clarified as cardiac, infectious, renal, others, or unknown.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill 2012 criteria of ANCA associated vasculitis and agree to sign informed consent

Exclusion Criteria:

* Do not agree to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled all the AAV patients that fulfill 2012 criteria of ANCA associated vasculitis and agree to sign informed
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Death | from date of baseline examination until the date of death from any cause, up to 60 months
  death from any cause
End stage renal disease or significant loss of renal function | from date of baseline examination until the date of first documented end stage renal disease or date of death from any cause, whichever came first, up to 60 months
  start of chronic dialysis or renal transplantation or irreversible development of glomerular filtration rate <15 ml/minute per 1.73m(2)

SECONDARY OUTCOMES:
Disease activity | Five years
  assessed by the proportion of patients with severe flares
Adverse events | Five years
  a. deaths (from all causes); b. grade 3 or higher infections; c. malignant conditions; d. venous thromboembolic events; e. cardiovascular events; f. hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Xiao, doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya hospital, Changsha, Hunan, China